CLINICAL TRIAL: NCT06092606
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial on DH001 Tablets in the Prevention of Doxorubicin-induced Cardiotoxicity in Cancer Patients
Brief Title: A Multicenter Clinical Trial on DH001 Tablets in the Prevention of Doxorubicin-induced Cardiotoxicity in Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monyan Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTR20232122
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Heart Failure; Arrhythmia; Doxorubicin Induced Cardiomyopathy; Doxorubicin Adverse Reaction
MeSH Terms: conditions — Neoplasms; Heart Failure; Arrhythmias, Cardiac | interventions — Control Groups; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group:DH001 placebo (Placebo Comparator): Medication: Once per day on an empty stomach in the morning. Treatment cycle: 3 days before the first administration of doxorubicin to the entire treatment cycle of doxorubicin.
  Dosage: DH001 placebo (8 tablets)
  Interventions: Drug: Control group:DH001 placebo
- Trial group: DH001 low-dose group (Experimental): Medication: once per day on an empty stomach in the morning. Treatment cycle: 3 days before the first administration of doxorubicin to the entire treatment cycle of doxorubicin.
  Dosage: DH001 200mg (4 tablets) + DH001 placebo (4 tablets)
  Interventions: Drug: Trial group: DH001 low-dose group
- Trial group: DH001 high-dose group (Experimental): Medication: Once per day on an empty stomach in the morning. Treatment cycle: 3 days before the first administration of doxorubicin to the entire treatment cycle of doxorubicin.
  Dosage: DH001 400mg (8 tablets).
  Interventions: Drug: Trial group: DH001 high-dose group

INTERVENTIONS:
Drug: Control group:DH001 placebo — Dosage: DH001 placebo (8 tablets)
  Other Names: Control group
  Arms: Control group:DH001 placebo
Drug: Trial group: DH001 low-dose group — Dosage: DH001 200mg (4 tablets) + DH001 placebo (4 tablets)
  Arms: Trial group: DH001 low-dose group
Drug: Trial group: DH001 high-dose group — Dosage: DH001 400mg (8 tablets).
  Arms: Trial group: DH001 high-dose group

SUMMARY:
Purpose：1. Preliminary evaluation of the preventive effect of DH001 on doxorubicin-induced cardiotoxicity in cancer patients 2.To explore appropriate dosages to provide basis for dosages in subsequent confirmatory studies 3.To evaluate the effect of DH001 on the efficacy of doxorubicin treatment in cancer patients 4.To evaluate the safety of DH001 in cancer patients treated with doxorubicin

DETAILED DESCRIPTION:
After the subjects sign the informed consent form, meet the inclusion criteria and do not meet the exclusion criteria, they will receive a random number according to the order of enrollment, and will be randomly assigned to the DH001 low-dose group (200 mg), DH001 high-dose group (400 mg) and control group in a 1:1:1 manner according to the randomization plan；Stratification factor: Patient's tumor type [lymphoma and non-lymphoma (breast cancer, soft tissue sarcoma, etc.)].

ELIGIBILITY:
Inclusion Criteria:

- Subjects who meet all the following criteria can be included in this study：

1. Newly diagnosed lymphoma or non-lymphoma patients (breast cancer, soft tissue sarcoma, etc.) as well as lymphoma or non-lymphoma patients that do not have a history of anthracycline treatment (doxorubicin, epirubicin, pyrandoxorubicin, daunorubicin, demethoxydaunorubicin, aclarithromycin, mitoxantrone, etc.)；Cancer patients should meet the following requirements:

1. Lymphoma：

   1. Lymphoma patients confirmed by histopathology；
   2. No previous history of anthracyclines treatment；
   3. Doxorubicin treatment planned for no less than 6 cycles；
2. Non-lymphoma (breast cancer, soft tissue sarcoma, etc.)：

   1. Subjects with malignant tumors (breast cancer, soft tissue sarcoma, etc.) confirmed by histopathology and/or cytology；
   2. Subjects planned to be treated with doxorubicin continuously for no less than 4 cycles（The cumulative dose of doxorubicin is no less than 240 mg/m2.）；
   3. Subjects with no history of systemic chemotherapy involving anthracyclines； 2.Age 18-75 years old, male or female； 3.ECOG PS score 0-1； 4.Expected survival ≥24 weeks； 5. Vital organs function well, that is, relevant examination indicators within 14 days before randomization meet the following requirements：

<!-- -->

1. Blood routine tests：

   1. Hemoglobin ≥95 g/L (no blood transfusion within 14 days)；
   2. Neutrophil count ≥1.5×109/L；
   3. Platelet count ≥75×109/L；
2. Blood biochemical tests：

   1. Total bilirubin ≤ 1.5×ULN ( upper limit of normal )；
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3.0×ULN；
   3. Creatinine (Cr) ≤1.5×ULN or creatinine clearance rate ≥ 60 ml/min (CockcroftGault formula)； 6.Male or female patients of childbearing potential who are willing to use effective contraceptive methods during the study, as well as within 6 months after the last dose of treatment (e.g., double barrier, condoms, oral or injectable contraceptives, intrauterine devices, etc.). All female patients will be considered to be of childbearing potential unless the female patient has undergone natural menopause, artificial menopause or sterilization (such as hysterectomy, bilateral adnexectomy or radioactive ovarian irradiation, etc.).The serum test results within 7 days prior to the enrollment of female patients must show that they are not pregnant , and they must be non-lactating.

      7.Subjects'participation should be voluntary，subjects have signed the informed consent form，show good compliance, and are able to actively cooperate with treatment and follow-up visits.

      Exclusion Criteria:

      - 1.Subjects scheduled to receive other anthracycline regimens； 2.Subjects who have previously received or plan to receive radiotherapy with a target area including the heart or left axillary lymph node； 3.HER-2 positive breast cancer patients； 4.Subjects with existing cardiac clinical symptoms or diseases that are not well controlled, such as：
      1. Cardiac Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) <55%；
      2. QTc > 450ms (men); QTc > 470ms (women) (QTc interval calculated using the Fridericia Formula; if QTc is abnormal, it can be detected three times continuously with an interval of 2 minutes, and the average value is then taken)；
      3. Serum biomarkers：

   <!-- -->

   1. Cardiac troponin T (cTnT, if applicable): cTnT > upper limit of normal ；
   2. cardiac troponin I（cTnI）：cTnI>upper limit of normal；
   3. N-terminal pro-BNP：NT-proBNP≥upper limit of normal；
   4. B-type natriuretic peptide（BNP，if applicable）：BNP≥upper limit of normal； 4）New York Heart Association Classification (NYHA standards) of cardiac function >Class II； 5） Unstable angina； 6） Heart failure； 7） Moderate valvular heart disease or above; 8） Myocardial infarction within 1 year before enrollment； 9）Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention； 5.Subjects with high blood pressure that is not well controlled using antihypertensive medication (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg) (based on the average of BP readings obtained from ≥2 measurements)，the above parameters are allowed to be achieved through the use of antihypertensive therapy；Subjects with a history of hypertensive crisis or hypertensive encephalopathy； 6.Subjects with type 1 diabetes（T1D）; 7.Subjects with a body mass index ≥28 kg/m2； 8.Subjects with a history of previous heart transplant or complex congenital heart disease.

      9.Subjects that have undergone major surgical treatment (except for diagnosis) within 4 weeks before enrollment or are expected to require major surgical treatment during the study period (except for tumor resection surgery)； 10.Subjects with congenital or acquired immunodeficiency diseases, including human immunodeficiency virus (HIV), or history of organ transplantation or allogeneic stem cell transplantation； 11.Subjects with known active infections or active pulmonary tuberculosis infections shall not be included in the study；However, patients infected with hepatitis B virus (HBV) and hepatitis C virus (HCV) whose condition is stable after antiviral treatment can be enrolled.

      12.Subjects with a history of other malignancies within 5 years, excluding adequately treated cervical cancer in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, and breast ductal carcinoma in situ.

      13.Subjects whom the investigators believe have lesions that require emergency palliative radiotherapy/emergency surgery (such as spinal cord compression, cerebral herniation, pathological fracture).

      14.Subjects possess physical examination or clinical experimental findings that, investigators believe, may interfere with the results or increase the subject's risk of treatment complications；subjects who suffer from other uncontrollable diseases.

      15.Subjects who are unable to swallow pills, subjects with malabsorption syndrome, or any condition that affects gastrointestinal absorption.

      16.Subjects with obvious mental disorders or epilepsy; subjects with no behavioral or cognitive abilities; drug addicts; pregnant or lactating women.

      17.Subjects who have participated in other clinical trials within 1 month before screening.

      18.Subjects determined unfit to participate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of cardiac events | 18-24 weeks
  The incidence of cardiac events in subjects during doxorubicin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Principal Investigator — Peking University Cancer Hospital & Institute; Hongmei Jing, Principal Investigator — Peking University Third Hospital; Hui Zhou, Principal Investigator — Hunan Cancer Hospital; Yufu Li, Principal Investigator — Henan Cancer Hospital; Hesheng He, Principal Investigator — The First Affilaited Hospital of Wannan Medical College; Zeping Zhou, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University; Wenbin Qian, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Xiaojia Wang, Principal Investigator — Zhejiang Cancer Hospital; Jiwei Liu, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Zhenchang Sun, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Harbin Institute of Hematology and Cancer, Harbin, Heilongjiang, China